CLINICAL TRIAL: NCT01650259
Title: Post Marketing Surveillance on Long Term Drug Use of Trazenta® Tablets in Patients With Type 2 Diabetes Mellitus
Brief Title: Long-term Daily Use of Trazenta® Tablets in Patients With Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 1218.95
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Results first posted 2019-05-10 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Oral antidiabetic drug (OAD)
  Interventions: Drug: OAD
- Trazenta
  Interventions: Drug: Trazenta

INTERVENTIONS:
Drug: OAD — OAD except Trazenta tablets
  Groups: Oral antidiabetic drug (OAD)
Drug: Trazenta — Linagliptin
  Groups: Trazenta

SUMMARY:
Study to investigate the safety and efficacy of long-term daily use of Trazenta® Tablets as monotherapy in patients with type 2 diabetes mellitus and to assess baseline characteristics of patients with type 2 diabetes mellitus starting Trazenta® Tablets or any other oral antidiabetic monotherapy (naïve or switched from prior therapy of different oral antidiabetic drug).

ELIGIBILITY:
Inclusion criteria:

* Male and female patients with type 2 Diabetes Mellitus who have never been treated with Trazenta tablets / Linagliptin (monotherapy) before enrollment. (Trazenta group)
* Patients with type 2 Diabetes Mellitus starting any other oral antidiabetic monotherapy (naïve or switched from prior therapy of different oral antidiabetic drug (OAD)) except Trazenta tablets. (OAD group)

Exclusion criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 3300
Sampling Method: Non-Probability Sample
Enrollment: 4876 (Actual)
Dates: Start 2012-07-23 (Actual); Primary Completion 2017-09-05 (Actual); Study Completion 2017-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- One Or Multiple Locations, Japan

REFERENCES:
- [Derived] Yabe D, Yamamoto F, Lund SS, Okamura T, Kadowaki T. Long-term safety and effectiveness of linagliptin by baseline body mass index in Japanese patients with type 2 diabetes: a 3-year post-marketing surveillance study. Expert Opin Drug Saf. 2022 Oct;21(10):1303-1313. doi: 10.1080/14740338.2022.2057948. Epub 2022 May 3. PMID 35418260
- [Derived] Yamamoto F, Ikeda R, Ochiai K, Hirase T, Hayashi N, Okamura T. Long-Term Safety and Effectiveness of Linagliptin in Japanese Patients with Type 2 Diabetes and Renal Dysfunction: a Post-Marketing Surveillance Study. Diabetes Ther. 2020 Feb;11(2):523-533. doi: 10.1007/s13300-019-00754-4. Epub 2020 Jan 13. PMID 31933070
- [Derived] Yamamoto F, Unno Y, Okamura T, Ikeda R, Ochiai K, Hayashi N. Long-Term Safety and Effectiveness of Linagliptin in Japanese Patients with Type 2 Diabetes Mellitus: A 3-Year Post-Marketing Surveillance Study. Diabetes Ther. 2020 Jan;11(1):107-117. doi: 10.1007/s13300-019-00723-x. Epub 2019 Nov 11. PMID 31713160

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this post marketing surveillance (PMS) study 4876 patients were registered: 2513 patients (Pts.) in Trazenta® Tablets group & 2363 patients in other Oral Antidiabetic Drug (OAD) group (grp). 2414 out of 2513 patients were treated (trt) with Trazenta® Tablets. For other OAD group only baseline data & no observation period.
Pre-assignment Details: Non-interventional,observational prospective study based on newly collected data under routine medical practice with 1 grp of Pts. treated with long-term daily use of Trazenta® Tablets for evaluation of baseline,safety& efficacy data & another grp of Pts. treated with any other oral antidiabetic monotherapy for collection of baseline data only.
Groups:
- Trazenta® Tablets: Patients with type 2 diabetes mellitus were administered orally with 5 milligram (mg) of Trazenta® tablets for 156 weeks or until discontinuation.
- Other OAD: Patients with type 2 diabetes mellitus who were treated with any other oral antidiabetic monotherapy except Trazenta® tablets
Period: Overall Study
Arm/Group | Trazenta® Tablets | Other OAD
Started | 2513 (Started are the registered patients) | 2363 (Started are the registered patients)
Completed | 1470 | 2128
Not Completed | 1043 | 235
Not completed — Improvement | 105 | 0
Not completed — Adverse Event | 127 | 0
Not completed — Lack of Efficacy | 143 | 0
Not completed — Lost to Follow-up | 435 | 0
Not completed — Patients had no visit after entry | 70 | 0
Not completed — CRF not collected | 98 | 82
Not completed — Not treated | 1 | 7
Not completed — Other than listed | 64 | 146

BASELINE CHARACTERISTICS:
Population: Baseline (bl) set: This set included all pts. of safety set for Trazenta tablets grp excluding pts. who were not diagnosed as type 2 diabetes mellitus or had important protocol violations (PV) with respect to treatments at bl. Pts. in other OAD grp were evaluated only for patient demographic & bl characteristics, excluding pts had important PV.
Groups:
- Total: Total of all reporting groups
Arm/Group | Trazenta® Tablets | Other OAD | Total
Number analyzed (Participants) | 2233 | 2128 | 4361
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at the time of start taking Trazenta® Tablets or other OAD is presented Population: SS
  Years | 66.7 (12.5) | 65.3 (12.6) | 66.0 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Number of patients is categorized as Male or Female. Population: SS
  Participants
    Female | 929 | 910 | 1839
    Male | 1304 | 1218 | 2522
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Race and Ethnicity were not collected in this trial. Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Drug Reactions (ADRs)
Description: An adverse drug reactions (ADR) was defined as an adverse event (AE) if either the investigator or the sponsor (or both) assessed the causal relationship of Trazenta® Tablets either as "Yes", "Probably yes" or "Can't be denied".
Time Frame: From start of the treatment until the end of this PMS, i.e. up to week 156
Population: Safety Set (SS): SS includes all patients who had received treatment of Trazenta® Tablets as mono therapy except those who were found to have no observation after enrolment, invalid registration, or invalid contract.
Measure: Number; unit: Percentage of Participants
Arm/Group | Trazenta® Tablets
Number analyzed (Participants) | 2235
Percentage of Participants | 10.74

2. Secondary Outcome: Change From Baseline in HbA1c at the Last Observation During the Observation Period.
Description: Change from baseline in Haemoglobin A1c (HbA1c) at the last observation during the observation period is presented as mean change from baseline and standard deviation (SD).
Time Frame: Baseline and 156 week or last observation
Population: Efficacy Set: A subset of the safety set, which includes all patients in the "safety set" except those who had no available efficacy data and/or who did not suffer from type 2 diabetes mellitus from the safety set.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Trazenta® Tablets
Number analyzed (Participants) | 2235
percentage of HbA1c | -0.67 (1.27)

ADVERSE EVENTS:
Time Frame: From first drug administration patient was observed until 156 weeks, up to 241 weeks.
Description: Safety Set (SS) (SS includes all patients who had received treatment of Trazenta® Tablets as mono therapy except those who were found to have no observation after enrolment, invalid registration, or invalid contract.) was used for adverse event reporting.
Arm/Group | Trazenta® Tablets
All-Cause Mortality (participants affected / at risk) | 34/2235
Serious Adverse Events (participants affected / at risk) | 116/2235
Other Adverse Events (participants affected / at risk) | 0/2235
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trazenta® Tablets (N=2235)
Pneumonia (Infections and infestations) | 3
Herpes zoster (Infections and infestations) | 2
Bacterial infection (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Polycythaemia (Blood and lymphatic system disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Alcoholism (Psychiatric disorders) | 1
Cerebral infarction (Nervous system disorders) | 12
Dementia (Nervous system disorders) | 5
Altered state of consciousness (Nervous system disorders) | 1
Carotid artery occlusion (Nervous system disorders) | 1
Dementia Alzheimer's type (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Parkinson's disease (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Cataract (Eye disorders) | 1
Cardiac failure (Cardiac disorders) | 4
Myocardial infarction (Cardiac disorders) | 4
Angina pectoris (Cardiac disorders) | 3
Angina unstable (Cardiac disorders) | 3
Acute myocardial infarction (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Prinzmetal angina (Cardiac disorders) | 1
Aortic dissection (Vascular disorders) | 1
Circulatory collapse (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Peripheral artery occlusion (Vascular disorders) | 1
Shock (Vascular disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Ileus (Gastrointestinal disorders) | 2
Enterocolitis (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Mechanical ileus (Gastrointestinal disorders) | 1
Bile duct stenosis (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hepatitis acute (Hepatobiliary disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Still's disease (Musculoskeletal and connective tissue disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 4
Acute kidney injury (Renal and urinary disorders) | 3
Renal impairment (Renal and urinary disorders) | 2
Death (General disorders) | 4
Sudden death (General disorders) | 2
Sudden cardiac death (General disorders) | 1
Biopsy liver (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood urea increased (Investigations) | 1
Blood uric acid increased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 2
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Patella fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1

LIMITATIONS AND CAVEATS:
The study was conducted in an unblinded manner and without controls. The explanatory power of the study results was limited and the study results should be interpreted with the necessary caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2013-04-04): https://cdn.clinicaltrials.gov/large-docs/59/NCT01650259/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-14): https://cdn.clinicaltrials.gov/large-docs/59/NCT01650259/SAP_001.pdf